CLINICAL TRIAL: NCT04953663
Title: A Multicenter, Blind, Randomized, Placebo-controlled Phase I / IIA Study to Evaluate the Safety, Tolerability, and Initial Efficacy of a Single Injection of Ischemia Tolerant Human Allogeneic Bone Marrow Mesenchymal Stem Cells in Patients With Ischemic Stroke
Brief Title: Clinical Plan of Ischemic Stroke
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2020093
Record Dates: First submitted 2021-06-27; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: 3 arms for phase 1, and 3 arms for pashe 2
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low dose group (Experimental): 0.5 × 10 ^ 6 / kg (body weight) of it-hMSC per person
  Interventions: Biological: it-hMSC
- Middle dose group (Experimental): 1 × 10 ^ 6 / kg (body weight) of it-hMSC per person
  Interventions: Biological: it-hMSC
- High dose group (Experimental): 2 × 10 ^ 6 / kg (body weight) of it-hMSC per person
  Interventions: Biological: it-hMSC
- Highest dose cell group (Experimental): Highest dose of it-hMSC
  Interventions: Biological: it-hMSC
- Sub high dose cell group (Experimental): Sub high dose of it-hMSC
  Interventions: Biological: it-hMSC
- placebo group (Placebo Comparator): placebo
  Interventions: Biological: it-hMSC

INTERVENTIONS:
Biological: it-hMSC — Different doses of it-hMSC

SUMMARY:
Stroke is the main cause of adult health damage. 20% of stroke survivors need institutional care after 3 months, and up to 30% of them have severe or permanent disability. Stem cells are a kind of pluripotent cells with the ability of self replication. The self-renewal and differentiation characteristics of mesenchymal stem cells, as well as cytokine secretion effect and immune characteristics, provide the possibility for mesenchymal stem cells to treat ischemic stroke. After the infusion of mesenchymal stem cells, the secretion of soluble media including growth factors and cytokines may be the main mechanism of mesenchymal stem cells.

DETAILED DESCRIPTION:
Stroke is the main cause of adult health damage. 20% of stroke survivors need institutional care after 3 months, and up to 30% of them have severe or permanent disability. Stem cells are a kind of pluripotent cells with the ability of self replication. The self-renewal and differentiation characteristics of mesenchymal stem cells, as well as cytokine secretion effect and immune characteristics, provide the possibility for mesenchymal stem cells to treat ischemic stroke. After the infusion of mesenchymal stem cells, the secretion of soluble media including growth factors and cytokines may be the main mechanism of mesenchymal stem cells. The main purpose of this study was to evaluate the safety and tolerance of intravenous injection of ischemia tolerant human allogeneic bone marrow mesenchymal stem cells in patients with ischemic stroke. The secondary objective was to evaluate the clinical efficacy of ischemic tolerant human allogeneic bone marrow mesenchymal stem cells in the treatment of ischemic stroke patients with neurological dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ≥ 18 years old;
2. The history showed that the last clinical diagnosis of ischemic stroke was more than 6 months;
3. The results of MRI at the first diagnosis and at the time of selection indicated that there was ischemic stroke and dysfunction;
4. There was no significant improvement in neurological function or functional defect 2 months before the study;
5. There is serious neurological dysfunction related to the diagnosis in Article 2, which leads to the subjects need the assistance of others to walk, or cannot complete the general activities of daily living independently;
6. NIHSS score was 6-20;
7. The life expectancy is more than 12 months;
8. Before treatment, the patient received standard medical care for secondary prevention of ischemic stroke, including but not limited to appropriate blood pressure and cholesterol control measures, use of antiplatelet drugs or anticoagulants (except prohibited cases);
9. Be able to understand and provide the signed informed consent, or ask the designated legal guardian or spouse to make the above decision voluntarily on behalf of the subjects;
10. It is reasonable to expect that patients will receive standard medical care for secondary prevention of ischemic stroke and participate in safety follow-up of all plans;
11. Organ function determined according to the following criteria:

Serum AST ≤ 2.5 × Upper normal limit (ULN);

Serum alanine aminotransferase (ALT) ≤ 2.5 × Normal upper limit;

Total serum bilirubin ≤ 1.5 × Normal upper limit;

In subjects without antithrombotic therapy, prothrombin time (PT) and partial thrombokinase time (PTT) ≤ 1.25 × Normal upper limit;

Serum albumin ≥ 3.0g/dl;

Absolute neutrophil count (ANC) ≥ 1500/ μ L；

Platelets ≥ 150000/ μ L；

Hemoglobin ≥ 9.0g/dl;

Serum creatinine ≤ 1.5 × Normal upper limit;

Serum amylase or lipase were in normal range.

Exclusion Criteria:

1. History of epilepsy;
2. History of tumor;
3. History of brain tumor and brain trauma;
4. hepatitis B, five surface antigens, e antigens, e antibodies and core antibodies were positive for any one, positive for hepatitis C virus antibody, positive for syphilis serum antibody or HIV positive.
5. Myocardial infarction occurred within 6 months before the trial;
6. Suffering from any other medical disease with clinical significance, or with abnormal mental or laboratory results, the researcher or the sponsor determines that participating in the trial will bring safety risks to the subjects;
7. Imaging examination showed subarachnoid hemorrhage or intracerebral hemorrhage in the past 12 months;
8. Participate in another study on the use of test drug or equipment within 3 months before treatment;
9. Participated in other stem cell therapy related research;
10. History of drug or alcohol abuse in the past year;
11. Women who are known to be pregnant, breast-feeding or have a positive pregnancy test (to be tested during the screening process) or plan to be pregnant during the trial;
12. Allergic to cattle and pork products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events rate | In 12 months
  Safety and tolerability of it-hMSC treatment
Rate of clinical significant changes in laboratory | In 12 months
  Safety and tolerability of it-hMSC treatment
Rate of abnormal neurological physical examination results | In 12 months
  Safety and tolerability of it-hMSC treatment
Rate of imaging changes | In 12 months
  Safety and tolerability of it-hMSC treatment

SECONDARY OUTCOMES:
Change of NIHSS scores | 1、3、6、9、12 months after treatment
  The improvement of neurological function was evaluated by neurological
Change of BI scores | 1、3、6、9、12 months after treatment
  The improvement of neurological function was evaluated by neurological
Change of mRS scores | 1、3、6、9、12 months after treatment
  The improvement of neurological function was evaluated by neurological
Change of MMSE scores | 1、3、6、9、12 months after treatment
  The improvement of neurological function was evaluated by neurological
Change of GDS scores | 1、3、6、9、12 months after treatment
  The improvement of neurological function was evaluated by neurological

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijin, China

IPD SHARING:
Plan to Share IPD: No